CLINICAL TRIAL: NCT04977778
Title: Effectiveness in Dental Plaque Reduction of Two Mouthwashes Containing Fatty Acids Compounds (F.A.G.) or Stannous Fluoride: a Comparative Study
Brief Title: Effectiveness in Dental Plaque Reduction of Mouthwashes Containing Fatty Acids Compounds (F.A.G.) or Stannous Fluoride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Davide Pietropaoli, PI, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 77593/2021
Record Dates: First submitted 2021-07-12; First posted 2021-07-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Gingivitis; Gingival Diseases
MeSH Terms: conditions — Gingivitis; Gingival Diseases | interventions — Mouthwashes; Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fatty Acids Compounds (FAG) (Active Comparator): Individuals taking FAG mouthwash
  Interventions: Drug: Fatty Acids Compounds (F.A.G.) Mouthwash
- Stannous Fluoride (SF) (Active Comparator): Individuals taking SF mouthwash
  Interventions: Drug: Stannous Fluoride (SF) Mouthwash

INTERVENTIONS:
Drug: Fatty Acids Compounds (F.A.G.) Mouthwash — Fatty Acids Compounds (F.A.G.) Mouthwash
  Arms: Fatty Acids Compounds (FAG)
Drug: Stannous Fluoride (SF) Mouthwash — Stannous Fluoride (SF) Mouthwash
  Arms: Stannous Fluoride (SF)

SUMMARY:
Comparative study on the efficacy of two mouthwashes Containing Fatty Acids Compounds (F.A.G.) or Stannous Fluoride in the reduction of plaque score in individuals with spontaneous gengivitis

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Smoking
* Drugs prior month
* Dental hygiene <6 months
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Change in plaque score | Baseline; 2 weeks
  Visual quantification of dental plaque amount on teeth buccal surfaces (wisdom teeth excluded).
  0% = no visible plaque on teeth surfaces 100% = plaque visible on all teeth surfaces

SECONDARY OUTCOMES:
Bleeding on Probing | Baseline; 2 weeks
  Quantifying gingival bleeding after gentle gum manipulation assessed on 6 points per tooth (exluded wisdom teeth).
  0% = No bleeding on all assessed points 100% = Bleeding on all assessed points

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, L’Aquila, IT, Italy

IPD SHARING:
Plan to Share IPD: Undecided